CLINICAL TRIAL: NCT06495008
Title: Taste and Smell Dysfunction in Patients More Than Two Years After Start of Immune Checkpoint Inhibitor Therapy
Acronym: TasteSPICIER
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 11303
Record Dates: First submitted 2024-01-02; First posted 2024-07-10 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Melanoma; Non-small Cell Lung Cancer (NSCLC); Urogenital Cancers
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Urogenital Neoplasms | interventions — Taste

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with cancer having finished immunotherapy >2 yrs ago
  Interventions: Other: no intervention, only questionnaires, saliva collection and taste/smell tests
- caregivers: Caregivers of patients with cancer
  Interventions: Other: no intervention, only questionnaires, saliva collection and taste/smell tests

INTERVENTIONS:
Other: no intervention, only questionnaires, saliva collection and taste/smell tests — no intervention, only questionnaires, saliva collection and taste/smell tests

SUMMARY:
Background of the study:

Immune checkpoint inhibitors (ICIs) are widely used as treatment for multiple cancer types and the number of patients with longterm disease control after ICIs is increasing. However, the use of ICIs is associated with adverse events (AEs) which can have a negative impact on quality of life (QoL). These AEs include oral manifestations, like alterations in taste and smell, xerostomia, and oral mucosal disorders, and could lead to unwanted weight loss. However, the characteristics of taste and smell dysfunction and xerostomia after treatment with ICIs are unknown. More insight in this phenomenon should be gained to make health care professionals aware of this problem to help patients cope with these AEs.

Objective of the study:

To determine the prevalence of taste and smell dysfunction in patients more than two years after ICI therapy - compared with a control group of caregivers.

Secondary objective: to assess the association between taste and smell dysfunction, and saliva secretion rate, saliva composition (pH, electrolyte and protein composition) and subjective feeling of a dry mouth (xerostomia) in patients more than two years after start of ICI therapy - compared with a control group of caregivers.

Study design:

Observational cross-sectional study.

Study population:

Patients (aged >18 years) with melanoma, non-small cell lung cancer (NSCLC) or urogenital cancers who have finished treatment with an ICI (CTLA-4 inhibitor, PD-(L)1 inhibitor, or both) >2 years ago, and their caregivers.

Primary study parameters/outcome of the study:

Taste and smell dysfunction, measured using taste strips and Sniffin' Sticks.

Secondary study parameters/outcome of the study:

Salivary flow rate, salivary pH, proteins and electrolytes, xerostomia, and perceived taste and smell dysfunction and impact of taste and smell dysfunction.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness (if applicable):

Participation in the study will include one study visit of approximately 1,5 hours. If possible, the study visit will be combined with a regular follow-up visit. In this study, no invasive procedures will be performed.

DETAILED DESCRIPTION:
In this cross-sectional study, patients with melanoma, NSCLC or urogenital cancer ≥ 2 years following ICI therapy and their caregivers will be included. The investigators will include patients who have previously participated in the study "Quality of life, cognitive function, and physical fitness of patients surviving more than 2 years after immune checkpoint inhibitor therapy" and additional patients who are under control at the departments of Medical Oncology and Pulmonary Disease and did not participate in this previous study. A patient cohort of patients and caregivers has already been built and patients who have given permission to be approached for future research again will be invited for our study.

Patients can be approached in two ways: 1) Patients will be asked during an outpatient clinic appointment by their clinical doctor if they can be approached afterwards by the investigator. When permission is given, the investigator will explain the study design and give the patient and the caregiver both a letter. These letters explains the study design and includes an informed consent form, 2) Patients who do not have an outpatient clinic appointment in the near future will be sent the letter with the study design and the informed consent form. In this letter, each participant will be asked to invite their caregiver to participate in this study. For this, a separate letter directed at the caregiver will be sent to the participant. Patients and caregivers are asked to contact the investigator team if they are willing to participate. If the patient consents, a single appointment will be made during a regular follow-up visit to the outpatient clinic. If the caregiver consents too, an appointment will be made with both participants at the same time, if possible. Patients can participate alone if the caregiver is not willing to participate, and vice versa.

During this visit, if patients and caregivers have no questions regarding the study or the study information that was sent, they are first asked to sign the informed consent. Next, saliva will be collected, and taste, smell and dry mouth will be subjectively and objectively be measured. Afterwards, characteristics will be taken from the patients' electronic file, including age, gender, medical history and medication use. As the caregivers do not have a medical file, they are asked for these characteristics.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with melanoma, NSCLC or urogenital cancers > 2 years since treatment with at least one cycle of immune checkpoint inhibitor (CTLA-4 inhibitor, PD-(L)1 inhibitor, or both) within the Department of Medical Oncology or Pulmonary Oncology of the UMCG.
* 2. Age >18 years at time of immune checkpoint inhibitor treatment
* 3. Understand or abide to the study procedures
* 4. Have given informed consent

A caregiver must meet all of the following criteria:

* 1. Age >18 years
* 2. Understand or abide to the study

Exclusion Criteria:

* 1. As previous or subsequent therapies, only surgery and palliative radiotherapy is allowed (excluding radiotherapy in the head-neck and brain region)
* 2. Previous treatment in the past ten years for malignancy other than melanoma (excluding non-melanoma skin cancer, cervical intra-epithelial neoplasia (CIN) or carcinoma in situ of breast) (for patients: other than current malignancy)
* 3. History of ear-nose-throat disease or auto-immune disorder affecting taste, smell, mouth mucosa, or saliva production (for patients: before start ICI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients (aged >18 years) with melanoma, non-small cell lung cancer (NSCLC) or urogenital cancers who have finshed treatment with an ICI (CTLA-4 inhibitor, PD-(L)1 inhibitor, or both) > 2 years ago, and their caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Taste function, score of test with taste strips | during single hospital visit more than 2 years after anticancer immunotherapy treatment
  Taste function measured using taste strips in patients compared to caregivers, resulting in a score of 0-16 points with 16 being the best outcome.

SECONDARY OUTCOMES:
Salivary flow rate in mL/min | during single hospital visit more than 2 years after anticancer immunotherapy treatment
  Salivary flow rate, stimulated and unstimulated production of saliva in cup in 5 minutes, in mL/min
Perceived taste and smell dysfunction, as determined using a standardized questionnaire | during single hospital visit more than 2 years after anticancer immunotherapy treatment
  Perceived taste and smell dysfunction, as determined using a standardized questionnaire
Perceived xerostomia, using standardized questionnaire | during single hospital visit more than 2 years after anticancer immunotherapy treatment
  Perceived xerostomia, using standardized questionnaire
Smell function | during single hospital visit more than 2 years after anticancer immunotherapy treatment
  Smell function measured using Sniffin' Sticks in patients compared to caregivers, resulting in a score of 0-16.

CONTACTS AND LOCATIONS:
Overall Officials: J. J. de Haan, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT06495008/Prot_SAP_001.pdf